CLINICAL TRIAL: NCT02329652
Title: Multi-functional Neuroprosthetic System for Restoration of Motor Function in Spinal Cord Injury
Acronym: NNP-UE+T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Bryden (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Case Western Reserve University (Other); Congressionally Directed Medical Research Programs (U.S. Federal Agency); FDA Orphan Products Division (Unknown)
Responsible Party: Sponsor-Investigator, Anne Bryden, Principal Investigator, MetroHealth Medical Center
Organization: MetroHealth Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NNP-UE+T; U01NS069517 (NIH); UH2NS103863 (NIH); OPD #5409 (Other Grant/Funding Number: FDA Office of Orphan Products Development); CDMRP-SC090230 (Other: CDMRP)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries; Spinal Cord Injury at C5-C7 Level; Spinal Cord Injury Cervical; Spinal Cord Injury at C5-C7 Level With Complete Lesion; Spinal Cord Injury at C5-C7 Level With Incomplete Lesion
Keywords: Neuroprosthesis; Functional Electrical Stimulation; Grasp; Posture; Standing; Function; Recovery; Device; Stimulation; Implant; Reach; Independence; Activities of Daily Living
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention - implant neuroprosthesis (Experimental): Receives implanted networked neuroprosthetic system for hand, arm, and trunk function. Undergoes functional training and assessment.
  Interventions: Device: Networked Neuroprosthetic System for Grasp and Trunk

INTERVENTIONS:
Device: Networked Neuroprosthetic System for Grasp and Trunk — Receive implanted networked neuroprosthesis

SUMMARY:
This study is to evaluate the use of a fully implanted device for providing hand function, reach, and trunk function to individuals with cervical spinal cord injury.

Funding Sources:

FDA OOPD NIH NINDS

DETAILED DESCRIPTION:
The goal of this project is to restore these multiple functions to these individuals through a comprehensive neuroprosthetic approach that addresses the overall needs of the individual. This approach involves all aspects of the implementation, including the implanted technology, the surgical installation, and the outcomes assessment through a coordinated team approach in order to maximize the functional independence gained by the individual. With this system, we propose that individuals who have a mid-cervical-level spinal cord injury will regain control over multiple functions, including grasp, reach, bed mobility, seated posture, restoration of an effective cough and bladder function. This ambitious and exciting goal is made possible by the culmination of our research and clinical deployment of neuroprosthetic systems for spinal cord injured subjects over the past 30 years. We anticipate that this system will not only provide increased independence in each of the targeted body functions, but will provide enough of an overall benefit to demonstrate significant improvements in quality of life and health outcomes.

In clinical feasibility studies with spinal cord injured subjects, our clinical research teams have demonstrated the control of bilateral hand function, bed mobility, postural control, restoration of an effective cough, and bladder control using chronically implanted neuroprostheses. Outcomes from each clinical study demonstrate that each system provides increased functional independence to the individual. Initially, only a single type of implanted system was implemented in any one individual, resulting in restoration of a single bodily function. Thus, it has been necessary for subjects to choose between available functions and select only one, despite the fact that each subject had multiple disabilities. In the past few years, we have progressed to implementing a few subjects with more than one system, such as providing both hand function and trunk stability. However, the fundamental limitation of the current approach has been technological; i.e. each implanted system is completely independent (both technically and programmatically), requiring separate technology to be developed for each function, and these systems are implemented by separate teams in separate surgical procedures. Thus, to this point, it has not been possible to address each individual's comprehensive needs and tailor an overall approach that maximizes their functional gains.

The proposed approach depends on the availability of a foundational platform technology that is capable of meeting our broad specifications. We have now achieved this milestone under separate funding, creating a revolutionary new implantable neuroprosthetic technology that is fully capable of providing the necessary technological base for our proposed research. This system, the Networked Neuroprosthetic System (NNPS), is a modular, scalable, and configurable network of fully implanted, networked modules capable of meeting or exceeding the needs of all of these neuroprosthetic applications. The NNPS provides a foundation which enables efficient technical refinements that optimize implementation of the system for each targeted application. The NNPS technology is currently operational and is undergoing fabrication and testing in preparation for final pre-clinical studies and human implantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical level spinal cord injury, either complete or incomplete; International Standards for Neurological Classification of Spinal Cord Injury (INCSCI) motor level of C4 through C8; American Spinal Injury Impairment Scale (AIS) grade A, B, C, or D; six months or more post-injury
* Biceps/brachialis/brachioradialis strength of 2/5 or higher on Manual Muscle Test
* Peripheral nerve innervation to upper extremity and trunk muscles, including a grade 3/5 or higher stimulated strength (Manual Muscle Test) in at least two of the following muscles in one arm: adductor pollicis, abductor pollicis brevis, flexor pollicis longus, extensor pollicis longus, extensor digitorum communis, flexor digitorum superficialis, flexor digitorum profundus, pronator quadratus, extensor carpi ulnaris, extensor carpi radialis brevis, extensor radialis longus, flexor carpi ulnaris, flexor carpi radialis, first dorsal interosseous; and in at least two of the following muscles: left/right gluteus maximus, left/right erector spinae, left/right quadratus lumborum,
* Age > 16 years
* Medically stable - cleared for surgery
* Able and willing to take part in study

Exclusion Criteria:

* Currently pregnant (neuroprosthesis implantation delayed until no longer pregnant)
* Other neurological conditions (multiple sclerosis, diabetes with peripheral nerve involvement)
* History of coagulopathy, HIV, severe cardiopulmonary disease, severe bradycardia, severe autonomic dysreflexia, or chronic obstructive pulmonary disease.
* Active untreated infection such as decubitus ulcer, urinary tract infection, pneumonia
* Presence of other active implantable medical devices with unknown or untested interaction with the NNP implant
* Active implantable medical device (AIMD) such as a pacemaker or defibrillator, with the exception of the implanted stimulator-telemeter (IST) or implanted receiver stimulator (IRS) systems developed by the Cleveland Functional Electrical Stimulation Center
* Unhealed fractures that prevent functional use of arm or trunk
* Less than six months post-injury (neuroprosthesis implantation delayed until criteria met)
* Extensive upper extremity denervation (fewer than two stimulatable hand muscles and two stimulatable trunk muscles)
* Involvement in other ongoing clinical studies that exclude concurrent until criteria met)
* Disorder or condition that require MRI monitoring
* Mechanical ventilator dependency
* Progressive SCI In subjects who are undergoing bilateral implantation, subjects should not have a history of autonomic dysreflexia, hypertension, diabetes or any condition which requires frequent blood pressure monitoring or frequent venipuncture.
* Adverse interaction between system components and typical electromagnetic (EM) sources in subject's home and work environments, including wheelchair or other active implantable devices.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Activities of Daily Living Abilities Test | Three months post-implant
  Evaluation of ability to perform activities of daily living when using the neuroprosthesis compared to ability when the neuroprosthesis is turned off.

SECONDARY OUTCOMES:
Grasp-Release Test | Pre-implant and three months post-implant
  Ability to pick up, move, and release six standard objects.

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ho CH, Triolo RJ, Elias AL, Kilgore KL, DiMarco AF, Bogie K, Vette AH, Audu ML, Kobetic R, Chang SR, Chan KM, Dukelow S, Bourbeau DJ, Brose SW, Gustafson KJ, Kiss ZH, Mushahwar VK. Functional electrical stimulation and spinal cord injury. Phys Med Rehabil Clin N Am. 2014 Aug;25(3):631-54, ix. doi: 10.1016/j.pmr.2014.05.001. PMID 25064792
- [Background] Peckham PH, Kilgore KL. Challenges and opportunities in restoring function after paralysis. IEEE Trans Biomed Eng. 2013 Mar;60(3):602-9. doi: 10.1109/TBME.2013.2245128. Epub 2013 Mar 7. PMID 23481680
- [Background] Makowski N, Campean A, Lambrecht J, Buckett J, Coburn J, Hart R, Miller M, Montague F, Crish T, Fu M, Kilgore K, Peckham PH, Smith B. Design and Testing of Stimulation and Myoelectric Recording Modules in an Implanted Distributed Neuroprosthetic System. IEEE Trans Biomed Circuits Syst. 2021 Apr;15(2):281-293. doi: 10.1109/TBCAS.2021.3066838. Epub 2021 May 25. PMID 33729949
- [Result] Kilgore KL, Hoyen HA, Bryden AM, Hart RL, Keith MW, Peckham PH. An implanted upper-extremity neuroprosthesis using myoelectric control. J Hand Surg Am. 2008 Apr;33(4):539-50. doi: 10.1016/j.jhsa.2008.01.007. PMID 18406958
- See also: Cleveland Functional Electrical Stimulation Center — http://fescenter.org